CLINICAL TRIAL: NCT06923826
Title: Sacituzumab Govitecan in Metastatic Salivary Gland and Thyroid Cancers (SG-SGTC) - A Phase 2 Multi-centre Trial
Brief Title: Sacituzumab Govitecan in Metastatic Salivary Gland and Thyroid Cancers (SG-SGTC)
Acronym: TROP2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECOS Ref. 2024-3605; CO-US-979-7131 (Other: Gilead)
Record Dates: First submitted 2025-03-12; First posted 2025-04-11 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2024-11

CONDITIONS: Salivary Gland Cancer; Thyroid Cancer
Keywords: salivary gland cancer; Sacituzumab govitecan; thyroid cancer
MeSH Terms: conditions — Salivary Gland Neoplasms; Thyroid Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Experimental): Participants with metastatic/ recurrent salivary gland cancers such as adenoid cystic carcinoma, mucoepidermoid carcinoma, adenocarcinoma NOS and salivary duct carcinoma.
  Each treatment cycle is 3 weeks. Treatment will be continued till disease progression, unacceptable toxicity or withdrawal of consent
  Interventions: Drug: Sacituzumab govitecan
- Cohort B (Experimental): Participants with metastatic/ recurrent well-differentiated or poorly differentiated radioactive iodine (RAI) refractory thyroid carcinoma. Each treatment cycle is 3 weeks. Treatment will be continued till disease progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Sacituzumab govitecan — Day 1 and Day 8: Sacituzumab Govitecan will be administered at the dose of 10 mg/kg via intravenous infusion.
  Other Names: Trodelvy

SUMMARY:
The goal of this clinical trial is to learn if the drug, sacituzumab govitecan, works to treat:

1. Salivary gland cancers that have spread to other parts of the body or come back after previous treatment, and cannot be removed by surgery
2. A type of thyroid cancer (specifically, differentiated thyroid carcinoma) that has spread to other parts of the body or come back after previous treatment, no longer responds to radioactive iodine treatment and cannot be removed by surgery

The main question it aims to answer is whether sacituzumab govitecan can treat the 2 conditions mentioned above in a safe and effective manner.

Participants will:

* Receive sacituzumab govitecan by intravenous (IV) infusion on Day 1 and Day 8 of each treatment cycle. Each treatment cycle is 21 days (3 weeks) long.
* Visit the clinic before each infusion for checkups and blood tests
* Go through CT/PET/MRI scan once every 6 weeks for the first 24 weeks, then every 9 weeks thereafter.
* Go through 2 tumour biopsies (if assessed by the doctor to be safe) at the start and at the end of study participation

Participants will continue to receive treatment with sacituzumab govitecan until their cancer stops responding to the drug or if they decide to withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

1. The participants (or legally acceptable representative if applicable) provide written consent for the trial.
2. At least 21 years of age on the day of signing informed consent.
3. Have histologically or cytologically confirmed diagnosis of advanced or unresectable salivary gland cancer or thyroid cancer, not amenable to local treatment.
4. Have measurable disease based on RECIST 1.1.
5. Patients with metastatic or recurrent unresectable advanced salivary gland cancers must have progressive disease within the previous 6 months and have seen at least 1 prior line of systemic treatment, unless the patients had contraindications to the systemic treatment considered standard of care or there was no standard of care for that particular salivary gland histological subtype.
6. Patients with unresectable metastatic or recurrent RAI refractory differentiated thyroid carcinoma, must have progressive disease within the previous 13 months and have seen at least 1 prior line of tyrosine kinase inhibitor (TKI), unless the patients had contraindications to the TKIs. Prior next generation sequencing is not mandated, but if known to harbour somatic pathogenic RET alteration or NTRK gene fusion, then the patient must have received 2 prior lines of TKIs, unless the patients had contraindications to the TKIs or declined the 2nd line of TKIs.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Have an adequate organ function. Specimens must be collected within 10 days prior to the start of study treatment.
9. Provision of blood and tumour tissue samples (newly obtained biopsy if clinically feasible or archival specimen) to support exploratory biomarker analysis.

Exclusion Criteria:

1. Has untreated brain metastases or leptomeningeal metastases.
2. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to first dose of study treatment.
3. Has received prior radiotherapy within 2 weeks of the start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
4. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
5. Known severe hypersensitivity reaction to Sacituzumab govitecan.
6. Has an active infection requiring systemic treatment. This includes TB (Bacillus Tuberculosis).
7. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
8. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
9. Recent cardiovascular thromboembolic event, such as the following:

   1. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤ 4 weeks before enrolment
   2. Symptomatic pulmonary embolism ≤ 4 weeks before enrolment
   3. Any history of acute myocardial infarction ≤ 6 months before enrolment
   4. Any history of heart failure meeting New York Heart Association (NYHA) Classification III or IV ≤ 6 months before enrolment
   5. Any event of ventricular arrhythmia ≥ Grade 2 in severity ≤ 6 months before enrolment
   6. Any history of cerebrovascular accident ≤ 6 months before enrolment
10. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial
11. A WOCBP who has a positive urine pregnancy test within 72 hours prior to first dose. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

    Note: In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative for subject to start receiving study medication.
12. Is not willing to practice contraception during the study, and for up to a period of at least 6 months after the last dose of SG:

    1. A woman of childbearing potential who does not agree to follow the contraceptive guidance on the use of effective contraception during the treatment period and for at least 6 months after the last dose of study medication.
    2. A male participant who does not agree to the use of effective contraception during the treatment period and for at least 3 months after the last dose of study treatment, and to refrain from donating sperm during this period.
13. History of having received a live virus vaccination (e.g., yellow fever, MMR, nasal flu, chicken pox or Zostavax) within 4 weeks prior to the first dose of trial treatment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  ORR is defined as the as the percentage of participants with a complete response (CR) or partial response (PR) according to response evaluation criteria in solid tumours (RECIST) version 1.1.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From date of treatment assignment until first documented progression or date of death, whichever occurs earlier, assessed up to 3 years
  PFS is defined as the time from treatment assignment to disease progression or death, whichever occurs first
Incidence of Treatment-Related Adverse Events (TRAEs) | From date of informed consent till 90 days following the date of last dose of study treatment.
  The frequency and outcome of TRAEs as assessed and graded according to the CTCAE version 5.0.
6-months Disease control rate (DCR) | Up to 6 months after initiating study treatment.
  6-months DCR is defined to be the percentage of participants with a complete response (CR), partial response (PR) or stable disease (SD) noted as the objective response status, according to RECIST version 1.1, at 6 months after initiating study treatment.
Correlation of ORR with Trop-2 expression in tumour samples | Up to 3 years
  Relationship between ORR and Trop-2 expression levels measured in tumour samples.

CONTACTS AND LOCATIONS:
Overall Officials: Wan Qin Dr Chong, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Cancer Institute Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Explain why IPD will not or might not be shared.

REFERENCES:
- [Background] Cubas R, Zhang S, Li M, Chen C, Yao Q. Trop2 expression contributes to tumor pathogenesis by activating the ERK MAPK pathway. Mol Cancer. 2010 Sep 21;9:253. doi: 10.1186/1476-4598-9-253. PMID 20858281
- [Background] Schlumberger M, Brose M, Elisei R, Leboulleux S, Luster M, Pitoia F, Pacini F. Definition and management of radioactive iodine-refractory differentiated thyroid cancer. Lancet Diabetes Endocrinol. 2014 May;2(5):356-8. doi: 10.1016/S2213-8587(13)70215-8. Epub 2014 Jan 30. No abstract available. PMID 24795243
- [Background] Shulin JH, Aizhen J, Kuo SM, Tan WB, Ngiam KY, Parameswaran R. Rising incidence of thyroid cancer in Singapore not solely due to micropapillary subtype. Ann R Coll Surg Engl. 2018 Apr;100(4):295-300. doi: 10.1308/rcsann.2018.0004. Epub 2018 Mar 15. PMID 29543059
- [Background] Mahmood U, Koshy M, Goloubeva O, Suntharalingam M. Adjuvant radiation therapy for high-grade and/or locally advanced major salivary gland tumors. Arch Otolaryngol Head Neck Surg. 2011 Oct;137(10):1025-30. doi: 10.1001/archoto.2011.158. PMID 22006781
- [Background] Licitra L, Cavina R, Grandi C, Palma SD, Guzzo M, Demicheli R, Molinari R. Cisplatin, doxorubicin and cyclophosphamide in advanced salivary gland carcinoma. A phase II trial of 22 patients. Ann Oncol. 1996 Aug;7(6):640-2. doi: 10.1093/oxfordjournals.annonc.a010684. PMID 8879381
- [Background] Guan H, Guo Z, Liang W, Li H, Wei G, Xu L, Xiao H, Li Y. Trop2 enhances invasion of thyroid cancer by inducing MMP2 through ERK and JNK pathways. BMC Cancer. 2017 Jul 14;17(1):486. doi: 10.1186/s12885-017-3475-2. PMID 28709407
- [Background] Rugo HS, Bardia A, Marme F, Cortes J, Schmid P, Loirat D, Tredan O, Ciruelos E, Dalenc F, Gomez Pardo P, Jhaveri KL, Delaney R, Valdez T, Wang H, Motwani M, Yoon OK, Verret W, Tolaney SM. Overall survival with sacituzumab govitecan in hormone receptor-positive and human epidermal growth factor receptor 2-negative metastatic breast cancer (TROPiCS-02): a randomised, open-label, multicentre, phase 3 trial. Lancet. 2023 Oct 21;402(10411):1423-1433. doi: 10.1016/S0140-6736(23)01245-X. Epub 2023 Aug 23. PMID 37633306
- [Background] Paz-Ares LG, Juan-Vidal O, Mountzios GS, Felip E, Reinmuth N, de Marinis F, Girard N, Patel VM, Takahama T, Owen SP, Reznick DM, Badin FB, Cicin I, Mekan S, Patel R, Zhang E, Karumanchi D, Garassino MC. Sacituzumab Govitecan Versus Docetaxel for Previously Treated Advanced or Metastatic Non-Small Cell Lung Cancer: The Randomized, Open-Label Phase III EVOKE-01 Study. J Clin Oncol. 2024 Aug 20;42(24):2860-2872. doi: 10.1200/JCO.24.00733. Epub 2024 May 31. PMID 38843511